CLINICAL TRIAL: NCT04454944
Title: Understanding Adoption of Clean Cookstoves
Brief Title: Understanding Adoption for Clean Cookstoves: A Demand Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Darby Jack, Associate Professor of Environmental Health Sciences, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: AAAS9921
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Consumer Behavior
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomized to 5 price levels and to 5 LPG cylinder exchange depots, for a total of 25 possible location/price combinations. Additionally, participants were enrolled into 4 arms (see arms description).
Masking Description: Prices and locations were public information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): All individuals in each arm will have a well-functioning LPG cookstove and gas cylinder. Participants in the control arm will receive no other intervention.
- No subsidy, distance variation (Experimental): All individuals in each arm will have a well-functioning LPG cookstove and gas cylinder. This intervention arm will receive an assigned depot where they have to make liquefied petroleum gas (LPG) purchases.
  Interventions: Behavioral: Distance allocation
- Subsidy, no distance variation (Experimental): All individuals in each arm will have a well-functioning LPG cookstove and gas cylinder. This intervention arm receives a price subsidy on liquefied petroleum gas (LPG) purchases.
  Interventions: Behavioral: LPG subsidy
- Subsidy, distance variation (Experimental): All individuals in each arm will have a well-functioning LPG cookstove and gas cylinder. This intervention arm receives a price subsidy on liquefied petroleum gas) (LPG) purchases an assigned depot where they have to make liquefied petroleum gas (LPG) purchases.
  Interventions: Behavioral: LPG subsidy; Behavioral: Distance allocation

INTERVENTIONS:
Behavioral: LPG subsidy — Different subsidy rates, ranging between 0% and 100% (listed below) will be written on cards. Individuals will randomly select a card to display the subsidy rate for each household. The card will be concealed with a scratch-off sticker, with a higher likelihood of drawing a high price (low subsidy) than a low price (high subsidy) given that take up will be higher in the latter group.
  Arms: Subsidy, distance variation; Subsidy, no distance variation
Behavioral: Distance allocation — We will set up fuel supply depots to increase the convenience and lower costs and hassle associated with traveling to an established filling station. The supply depots will mirror a recirculation model of LPG distribution currently being piloted by the National Petroleum Authority of Ghana. Households will be randomly assigned to one of the supply depots in advance or to continue refilling their cylinder at the filling station.
  Arms: No subsidy, distance variation; Subsidy, distance variation

SUMMARY:
The aim of the Adoption study is to determine how best to encourage people to adopt clean cookstoves in order to diminish the global health risk of household air pollution. The study harnesses an existing cohort in Ghana to study factors that increase the adoption of clean cookstoves, and to test strategies to promote adoption and continued use. Limited past research has shown that the demand for clean cookstoves is low, and that households continue to use traditional hearths even when they have clean cookstoves. This behavior threatens to undermine clean cookstove intervention programs, such as those promoted by the Global Alliance for Clean Cookstoves. The proposed study aims to ascertain the demand curve for liquified petroleum gas (LPG) in the Kintampo North Municipality and South district.

DETAILED DESCRIPTION:
The study will assess if demand for LPG in rural settings in Ghana is price elastic - and by how much - by providing different levels of LPG price subsidies. It will also ascertain if demand is influenced by distance by allocating participants to varying distances to points of LPG supply. Finally, it will assess factors that could affect the demand for LPG such as availability and price of other fuels for cooking, and income levels.

In particular the objectives of the study are:

1. To determine if demand for LPG is price elastic
2. To determine if demand for LPG is influenced by distance
3. To ascertain what other factors aside the price of LPG, and distance to point of LPG supply, determine the demand for LPG
4. To document the successes and challenges of introducing a subsidy for LPG in rural settings

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Primary cook of the household
* Part of the Ghana Randomized Air Pollution and Health Study (GRAPHS) sample or reside in a sample village
* Owns an LPG stove and cylinder (provided by the project in the case of newly recruited households)

Exclusion Criteria

- Temporarily residing in study area.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Demand for LPG | 6 months
  The primary outcome will be measured by the number of LPG cylinder purchases and/or refills by the study participant.

CONTACTS AND LOCATIONS:
Overall Officials: Darby Jack, PhD, Principal Investigator — Columbia University
Locations (2):
- Columbia University Medical Center, New York, New York, United States
- Kintampo Medical Research Center, Kintampo, Ghana

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared between the study teams at the Kintampo Health Research Center, Columbia University and University of California, Santa Barbara. This data will not include medical or clinical information.
  We plan to create a public use de-identified dataset that will be made available via the Ghana Open Data Initiative or a similar repository.
Supporting Information: Study Protocol, SAP, ICF